CLINICAL TRIAL: NCT01849263
Title: Phase 2 Trial of Single-Agent Ibrutinib (PCI-32765) in Relapsed or Refractory Follicular Lymphoma
Brief Title: Ibrutinib in Treating Patients With Relapsed or Refractory Follicular Lymphoma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2013-00887; NCI-2013-00887 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); MC1282; 9271 (Other: Mayo Clinic in Rochester); 9271 (Other: CTEP); N01CM00032 (NIH); N01CM00099 (NIH); P30CA015083 (NIH); U10CA180821 (NIH); NCT02989532 (obsolete NCT alias)
Record Dates: First submitted 2013-05-06; First posted 2013-05-08 (Estimated); Results first posted 2018-04-26 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Grade 3a Follicular Lymphoma; Recurrent Grade 1 Follicular Lymphoma; Recurrent Grade 2 Follicular Lymphoma; Recurrent Grade 3 Follicular Lymphoma; Refractory Follicular Lymphoma
MeSH Terms: conditions — Lymphoma, Follicular | interventions — ibrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (ibrutinib) (Experimental): Patients receive ibrutinib PO QD on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients with progressive disease at the end of course 2 may continue on therapy until the end of course 5 at the discretion of the treating physician.
  Interventions: Drug: Ibrutinib; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Drug: Ibrutinib — Given PO
  Other Names: BTK Inhibitor PCI-32765; CRA 032765; CRA-032765; CRA032765; Imbruvica; PCI 32765; PCI-32765; PCI32765
Other: Laboratory Biomarker Analysis — Correlative studies

SUMMARY:
This phase II trial studies how well ibrutinib works in treating patients with follicular lymphoma that has come back after a period of improvement or does not respond to treatment. Ibrutinib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Evaluate the overall response rate of ibrutinib in patients with relapsed or refractory follicular lymphoma.

SECONDARY OBJECTIVES:

I. Assess the safety and tolerability of ibrutinib in patients with follicular lymphoma.

II. Evaluate overall survival, time to response, duration of response, progression-free survival, time to treatment failure, and time to subsequent treatment.

TERTIARY OBJECTIVES:

I. Describe the relationship between interim positron emission tomography (PET)/computed tomography (CT) scan results, CT response, and response duration.

II. Biomarker studies including exploring associations between ibrutinib response and somatic mutations identified in follicular lymphoma, whole transcriptome shotgun sequencing (ribonucleic acid-sequencing [RNA-seq]), exploration of inhibition of Bruton's tyrosine kinase (BTK) and other kinases, expression of cytokines, chemokines, and other proteins with an aim to develop predictors of response and resistance.

III. Assess changes in various cancer-derived molecules in the blood over the course of treatment with ibrutinib.

IV. As part of ongoing research for Phase II Consortium (P2C) studies, we are banking paraffin-embedded tissue blocks/slides and blood products for future studies.

OUTLINE:

Patients receive ibrutinib orally (PO) once daily (QD) on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients with progressive disease at the end of course 2 may continue on therapy until the end of course 5 at the discretion of the treating physician.

After completion of study treatment, patients are followed up every 3 months until progressive disease, and then every 6 months for 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of follicular lymphoma, grade 1, 2, or 3a

  * Note: Fresh (frozen) tumor biopsy must be available or attempted; a frozen tumor biopsy equivalent to a minimum of four at least 16 gauge needle cores is an important component of this study; patients without adequate frozen material should have a biopsy performed to obtain material; if biopsy is performed and does not yield adequate material, the patient is still eligible for the study; if a biopsy cannot be done safely, the patient may still be eligible for the study if permission is granted in writing (email) by the study chair (Dr. Nancy Bartlett) or her designees; Dr. Bartlett may be consulted to discuss situations involving invasive biopsy procedures that may pose an increased risk to the patient
* Measurable disease as defined by a lymph node or tumor mass that is >= 1.5 cm in at least one dimension by CT or the CT portion of the PET/CT
* Relapsed or refractory follicular lymphoma which has progressed during or following 1 or more prior chemotherapy regimens for lymphoma
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0, 1 or 2
* Absolute neutrophil count >= 750/mm^3 (0.75 x 10^9/L)
* Hemoglobin >= 8.0 g/dL
* Platelets >= 30,000/mm^3 (30 x 10^9/L)
* Total bilirubin =< 1.5 x institutional upper limit of normal (ULN) unless Gilbert's syndrome or disease infiltration of the liver is present
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.0 x institutional ULN
* Creatinine =< 2.0 x institutional ULN
* Creatinine clearance (estimated [est.] glomerular filtration rate [GFR] Cockcroft-Gault) >= 30 mL/min
* Negative serum pregnancy test done =< 7 days prior to registration for women of childbearing potential only
* Ability to understand and the willingness to sign a written informed consent document
* Willingness to provide biologic samples for correlative research purposes

Exclusion Criteria:

* Any of the following:

  * Chemotherapy/systemic therapy =< 4 weeks prior to registration
  * Radiotherapy =< 4 weeks prior to registration
  * Nitrosoureas or mitomycin C =< 6 weeks prior to registration
  * Those who have not recovered from adverse events due to agents administered more than 4 weeks earlier
  * Major surgery =< 10 days prior to registration or minor surgery =< 7 days prior to registration
  * Prior therapy with ibrutinib or another Bruton's tyrosine kinase inhibitor
  * Receiving any other investigational agents
* Active central nervous system (CNS) involvement
* Receiving any medications or substances that are strong inhibitors or inducers of cytochrome P450 family 3 subfamily A member 4/5 (CYP3A4/5)
* Any of the following:

  * Pregnant women
  * Nursing women
  * Men or women of childbearing potential who are unwilling to employ adequate contraception

    * Note: Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation; should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately; men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 4 months after completion of ibrutinib administration
    * Note: Breastfeeding should be discontinued if the mother is treated with ibrutinib
* Human immunodeficiency virus (HIV)-positive patients on antiretroviral therapy are ineligible; appropriate studies will be undertaken in patients receiving combination antiretroviral therapy when indicated

  * Note: HIV-positive patients who are not on anti-viral medications that are strong CYP3A4/5 inhibitors and who do not have cluster of differentiation (CD)4 counts less than the lower limit of normal by institutional criteria are eligible; no patients with CD4 counts below institutional normals are eligible
* Known active infection with hepatitis C virus (HCV) or hepatitis B virus (HBV)
* Known histological transformation from follicular lymphoma to diffuse large B-cell lymphoma

  * Note: A prior history of adequately treated transformed lymphoma does not exclude a patient if the current active disease is biopsy-proven follicular lymphoma
* History of stroke or intracranial hemorrhage =< 6 months prior to the first dose of study drug
* Requires anticoagulation with warfarin or similar vitamin K antagonist

  * Note: Warfarin or similar vitamin K antagonist must have been discontinued at least 28 days prior to study entry
* Patient has the inability to swallow tablets
* Uncontrolled intercurrent illness including, but not limited to:

  * Ongoing or active infection,
  * Uncontrolled diabetes mellitus
  * Cardiac disease
  * Psychiatric illness/social situations that would limit compliance with study requirements
* "Currently active" second malignancy, other than non-melanoma skin cancers

  * Note: Patients are not considered to have a "currently active" malignancy if they have completed anti-cancer therapy, and are considered by their physician to be at less than 30% risk of relapse
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to ibrutinib
* Concurrent treatment with therapeutic doses (> 20 mg prednisone or equivalent) of systemic steroids within 14 days of start of protocol therapy
* Prior history of allogeneic stem cell transplant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2013-04-02 (Actual); Primary Completion 2016-06-03 (Actual); Study Completion 2026-03-19 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Nancy L Bartlett, Principal Investigator — Mayo Clinic
Locations (13):
- United States (8):
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Metro Minnesota Community Oncology Research Consortium, Saint Louis Park, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - University of Wisconsin Carbone Cancer Center - University Hospital, Madison, Wisconsin
- Canada (3):
  - Juravinski Cancer Centre at Hamilton Health Sciences, Hamilton, Ontario
  - Kingston Health Sciences Centre, Kingston, Ontario
  - University Health Network-Princess Margaret Hospital, Toronto, Ontario
- Singapore (2):
  - National University Hospital Singapore, Singapore
  - National Cancer Centre Singapore, Singapore

REFERENCES:
- [Derived] Bartlett NL, Costello BA, LaPlant BR, Ansell SM, Kuruvilla JG, Reeder CB, Thye LS, Anderson DM, Krysiak K, Ramirez C, Qi J, Siegel BA, Griffith M, Griffith OL, Gomez F, Fehniger TA. Single-agent ibrutinib in relapsed or refractory follicular lymphoma: a phase 2 consortium trial. Blood. 2018 Jan 11;131(2):182-190. doi: 10.1182/blood-2017-09-804641. Epub 2017 Oct 26. PMID 29074501

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Forty-one patients were enrolled to this study. One patient cancelled prior to beginning protocol treatment and was excluded from all analyses.
Groups:
- Treatment (Ibrutinib): Patients receive 560 mg ibrutinib PO QD on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients with progressive disease at the end of course 2 may continue on therapy until the end of course 5 at the discretion of the treating physician.
Period: Overall Study
Arm/Group | Treatment (Ibrutinib)
Started | 40
Completed | 40
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: All participants that started protocol treatment are included.
Arm/Group | Treatment (Ibrutinib)
Number analyzed (Participants) | 40
Age, Continuous [Median (Full Range); unit: years] | 64 [46 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 28
Region of Enrollment [Number; unit: participants]
  Canada | 5
  Singapore | 2
  United States | 33

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate
Description: Overall response rate defined as a partial response (PR) or complete response (CR) as the objective status at any time during treatment, evaluated using the Cheson et al. Revised Response Criteria for Malignant Lymphoma. Ninety-five percent binomial confidence intervals for the true success proportion will be calculated.
  A CR is defined as the disappearance of all evidence of disease. A PR is defined as ≥ 50% decrease in the sum of the products of dimensions (SPD) of up to 6 largest dominant masses; no increase in size of other nodes and regression on CT, and no increase in size of liver/spleen.
Time Frame: Up to 5 years
Population: All patients that began protocol treatment were included in this analysis.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Treatment (Ibrutinib)
Number analyzed (Participants) | 40
proportion of participants | 0.375 [0.227 to 0.542]

2. Secondary Outcome: Duration of Response
Description: Duration of response is defined as the time from first evidence of a response to the first documented time of progressive disease (PD). Response and Progression were assessed using the Cheson et al. Revised Response Criteria for Malignant Lymphoma. > > A CR is defined as the disappearance of all evidence of disease. A PR is defined as ≥ 50% decrease in the sum of the products of dimensions (SPD) of up to 6 largest dominant masses; no increase in size of other nodes and regression on CT, and no increase in size of liver/spleen.Estimated using the method of Kaplan-Meier.>
  > Progressive Disease (PD) is defined as any new lesion or increase by ≥ 50% of previously involved sites from nadir.
Time Frame: Time from the date at which the patient's objective status is first noted to be a CR or PR to the earliest date progression is documented, assessed up to 5 years
Population: All patients that reported a response during treatment are included in this analysis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Ibrutinib)
Number analyzed (Participants) | 15
months | 13.9 [5.8 to NA] — Too few events occurred to estimate the upper bound of the confidence interval.

3. Secondary Outcome: Overall Survival
Description: Overall Survival is defined as the time from registration to death due to any cause. Estimated using the method of Kaplan-Meier.
Time Frame: Assessed up to 5 years
Population: All patients beginning protocol treatment are included in this endpoint.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Ibrutinib)
Number analyzed (Participants) | 40
months | NA [NA to NA] — Too few events have occurred to estimate a median and confidence interval.

4. Secondary Outcome: Progression-free Survival
Description: Progression-Free Survival is defined as the time from registration to documented progression or death due to any cause, whichever occurs first. Estimated using the method of Kaplan-Meier.
Time Frame: Time from registration to progression or death due to any cause, assessed up to 5 years
Population: All patients beginning protocol treatment are included in this endpoint.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Ibrutinib)
Number analyzed (Participants) | 40
months | 14.0 [7.4 to 16.3]

5. Secondary Outcome: Time to Response
Description: Time to response is defined for all evaluable patients who have achieved a confirmed response as the time from the date of registration to the date at which the patient's objective status is first noted to be a CR or PR.The median and 95% confidence interval will be calculated using the methods of Kaplan-Meier.
Time Frame: Time from the date of registration to the date at which the patient's objective status is first noted to be a CR or PR, assessed up to 5 years
Population: All patients reporting a response during treatment are included in this analysis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Ibrutinib)
Number analyzed (Participants) | 15
months | 4.6 [1.8 to 10.4]

6. Secondary Outcome: Time to Subsequent Treatment
Description: Time to subsequent treatment is defined as the time from registration to the date of initiation of subsequent treatment for lymphoma. The distribution of time to subsequent treatment will be estimated using the method of Kaplan-Meier.
Time Frame: Time from registration to the date of initiation of subsequent treatment for lymphoma, assessed up to 5 years
Population: All patients beginning protocol treatment were included in this endpoint analysis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Ibrutinib)
Number analyzed (Participants) | 40
months | 17.7 [13.4 to 28.4]

7. Secondary Outcome: Time to Treatment Failure
Description: Time to treatment failure is defined as the time from registration to the date of treatment discontinuation due to any reason. The distribution of time to treatment failure will be estimated using the method of Kaplan-Meier.
Time Frame: Time from registration to the date of treatment discontinuation due to any reason, assessed up to 5 years
Population: All patients beginning protocol treatment were included in this endpoint analysis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Ibrutinib)
Number analyzed (Participants) | 40
months | 10.0 [6.0 to 16.2]

ADVERSE EVENTS:
Time Frame: Adverse events were collected at the end of each cycle of treatment, up to cycle 35.
Description: Adverse events were recorded at the end of each cycle of treatment.
Arm/Group | Treatment (Ibrutinib)
All-Cause Mortality (participants affected / at risk) | 1/40
Serious Adverse Events (participants affected / at risk) | 10/40
Other Adverse Events (participants affected / at risk) | 40/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Ibrutinib) (N=40)
Spleen disorder (Blood and lymphatic system disorders) | 1 (1)
Cardiac disorders - Other, specify (Cardiac disorders) | 1 (1)
Chest pain - cardiac (Cardiac disorders) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 2 (3)
Gastric hemorrhage (Gastrointestinal disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Infections and infestations - Other, specify (Infections and infestations) | 2 (2)
Lung infection (Infections and infestations) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1)
Hematoma (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Ibrutinib) (N=40)
Anemia (Blood and lymphatic system disorders) | 16 (62)
Leukocytosis (Blood and lymphatic system disorders) | 3 (3)
Cardiac disorders - Other, specify (Cardiac disorders) | 1 (1)
Ear and labyrinth disorders - Other, specify (Ear and labyrinth disorders) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 1 (1)
Blurred vision (Eye disorders) | 1 (1)
Cataract (Eye disorders) | 1 (1)
Conjunctivitis (Eye disorders) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 2 (3)
Bloating (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 6 (8)
Diarrhea (Gastrointestinal disorders) | 21 (130)
Dry mouth (Gastrointestinal disorders) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (3)
Flatulence (Gastrointestinal disorders) | 1 (1)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 2 (2)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 2 (4)
Hemorrhoidal hemorrhage (Gastrointestinal disorders) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 4 (15)
Nausea (Gastrointestinal disorders) | 13 (35)
Oral pain (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 8 (8)
Edema limbs (General disorders) | 6 (15)
Fatigue (General disorders) | 27 (145)
Fever (General disorders) | 2 (2)
Flu like symptoms (General disorders) | 2 (4)
Pain (General disorders) | 1 (1)
Bladder infection (Infections and infestations) | 1 (2)
Conjunctivitis infective (Infections and infestations) | 1 (1)
Gum infection (Infections and infestations) | 1 (2)
Infections and infestations - Other, specify (Infections and infestations) | 3 (3)
Lung infection (Infections and infestations) | 3 (4)
Otitis media (Infections and infestations) | 1 (1)
Sinusitis (Infections and infestations) | 4 (5)
Skin infection (Infections and infestations) | 2 (2)
Upper respiratory infection (Infections and infestations) | 7 (10)
Urinary tract infection (Infections and infestations) | 2 (2)
Vaginal infection (Infections and infestations) | 2 (2)
Bruising (Injury, poisoning and procedural complications) | 6 (12)
Alanine aminotransferase increased (Investigations) | 2 (3)
Alkaline phosphatase increased (Investigations) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 2 (4)
Blood bilirubin increased (Investigations) | 4 (6)
CD4 lymphocytes decreased (Investigations) | 1 (1)
Lymphocyte count decreased (Investigations) | 11 (52)
Neutrophil count decreased (Investigations) | 5 (16)
Platelet count decreased (Investigations) | 23 (137)
Weight loss (Investigations) | 1 (7)
White blood cell decreased (Investigations) | 5 (8)
Anorexia (Metabolism and nutrition disorders) | 3 (4)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (2)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1)
Hypernatremia (Metabolism and nutrition disorders) | 1 (2)
Hyperuricemia (Metabolism and nutrition disorders) | 2 (3)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (5)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (32)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Dizziness (Nervous system disorders) | 2 (2)
Dysgeusia (Nervous system disorders) | 3 (4)
Headache (Nervous system disorders) | 2 (4)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1)
Urinary tract obstruction (Renal and urinary disorders) | 1 (1)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (5)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (5)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (3)
Dry skin (Skin and subcutaneous tissue disorders) | 3 (8)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (2)
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 7 (16)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 5 (9)
Skin ulceration (Skin and subcutaneous tissue disorders) | 1 (1)
Hematoma (Vascular disorders) | 1 (4)
Hypertension (Vascular disorders) | 1 (2)
Thromboembolic event (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less